CLINICAL TRIAL: NCT02907931
Title: Carotid Doppler Ultrasound for the Measurement of Intravascular Volume Status During Lower Body Negative Pressure Simulation
Brief Title: Carotid Doppler Ultrasound for the Measurement of Intravascular Volume Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1608018234
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Hypotension; Sepsis
Keywords: hemodynamics; ultrasonography
MeSH Terms: conditions — Hypotension; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects (Experimental): Lower Body Negative Pressure
  Interventions: Other: Point of Care Ultrasound

INTERVENTIONS:
Other: Point of Care Ultrasound

SUMMARY:
Ultrasound represents an attractive non-invasive method to assess hemodynamic status. Understanding dynamic changes in hemodynamics in situations such as hypovolemia, sepsis, and cardiogenic shock can potentially help improve patient care. However, the inter-rater reliability and accuracy of how various ultrasound measurements reflect dynamic changes in physiology remains incompletely understood. Overall our aims are to investigate the use of ultrasound in a controlled setting, specifically using lower body negative pressure (LBNP), which can simulate hypovolemia at varied levels in human volunteers.

Aim 1: To determine the change in carotid blood flow (measured by velocity time integral, VTI) in subjects undergoing simulated hypovolemia at LBNP levels that precede vital sign changes.

Hypothesis: Carotid VTI will demonstrate significant changes that precede vital sign changes in simulated hypovolemia.

Aim 2: To compare transcranial color Doppler indices of cerebral blood flow with carotid blood flow, as assessed by VTI of the common carotid artery.

Hypothesis: Changes in transcranial color Doppler indices of cerebral blood flow will be mirrored by changes in carotid blood flow, indicating carotid VTI is an adequate surrogate for measuring cerebral blood flow in variable states of central hypovolemia. However, if cerebral blood flow remains more constant than carotid blood flow throughout varying levels of hypovolemia, our assumption is that cerebral autoregulation alters the relationship between carotid and cerebral blood flow. The more complex procedure of Transcranial Doppler ultrasound (TCD) must be performed to obtain valid assessments of cerebral blood flow.

DETAILED DESCRIPTION:
Study Design: This is a prospective laboratory study using human volunteers.

Study Setting and Subjects: The study will take place in The John B. Pierce Laboratory where volunteers will be subjected to lower body negative pressure using the on-site LBNP chamber.

Protocol: Study subjects will be instructed to refrain from caffeine, alcohol, or cigarettes within 12 hours of the protocol, but will otherwise be allowed their routine oral intake prior to enrollment. The chamber is constructed of a sealed wood and acrylic box that is connected to a vacuum. Subjects will be placed into the chamber, which is sealed to the level of their pelvis by a neoprene skirt. Chamber pressure is transduced to an electronic digital manometer. The pressure in the chamber will reduced rapidly and held for 15-minute intervals at -5, -10, -15, and -20 mm Hg. If the subject becomes lightheaded, nauseated, or does not tolerate the test run in any way; negative pressure will be stopped.

Subjects will be monitored with continuous electrocardiogram monitoring, a standard automated blood pressure cuff, and a noninvasive beat-to-beat hemodynamic monitor (Finometer, Finapres Medical Systems, Amsterdam, The Netherlands). All carotid ultrasound measurements will be performed by specifically trained emergency physicians, using a Philips ultrasound machine (Philips Medical Systems, Andover, MA) equipped with phased and linear array probes programmed with Doppler capability. For transcranial Doppler imaging, we will use a 5- to 1-MHz sector array transducer and an Iu-22 ultrasound system (Philips Healthcare, Best, the Netherlands). Duplex sonography will be performed at the lower end of the frequency range (1-2 MHz) for better sound wave penetration of selected bone windows. For both the common carotid artery and transcranial portion of this study, we will obtain spectral Doppler waveform tracings and record measurements of corresponding vessel diameters. We will use data generated from software analysis of these spectral tracings to calculate hemodynamic parameters of interest to our study. Calculations are based on Bernoulli's principles of fluid dynamics.

ELIGIBILITY:
Inclusion criteria:

1. Generally healthy
2. Able to provide informed consent
3. Over 18 years of age

Exclusion criteria:

1. Non-English speaking or decisionaly impaired
2. Significant medical illness (as determined by the study physician, JC)
3. Taking vasoactive medications
4. Older than 60 years of age
5. Inability to lie flat for prolonged period
6. Severe claustrophobia
7. Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-09; Primary Completion 2018-07 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
changes in carotid blood flow (measured by velocity time integral, VTI) in subjects undergoing simulated hypovolemia | over the course of 1-2 hours during which subjects will undergo incremental changes in lower body negative pressure
  We will attach adhesive electrodes to your chest which allow us to monitor and record your vital signs. You will lie on your back on a table with the lower half of your body enclosed in a box. The box has a vacuum that creates suction and causes blood to pool in your legs and feet. Next you will do a Lower Body Negative Pressure test. For this test, you will lie with your lower body in the box while we apply increasing levels of suction, over 4 different intervals, lasting 2 minutes each. We will repeat the suction for longer times at each interval and obtain ultrasound images of blood vessels in your head and neck. Each interval may last up to 20 minutes for a total of up to 80 minutes time spent in the chamber.

CONTACTS AND LOCATIONS:
Overall Officials: Jill C Crosby, MD, MHS, Principal Investigator — Yale University
Locations (1):
- John B. Pierce Laboratory, New Haven, Connecticut, United States

REFERENCES:
- [Background] Marik PE. Iatrogenic salt water drowning and the hazards of a high central venous pressure. Ann Intensive Care. 2014 Jun 21;4:21. doi: 10.1186/s13613-014-0021-0. eCollection 2014. PMID 25110606
- [Background] Marik PE, Levitov A, Young A, Andrews L. The use of bioreactance and carotid Doppler to determine volume responsiveness and blood flow redistribution following passive leg raising in hemodynamically unstable patients. Chest. 2013 Feb 1;143(2):364-370. doi: 10.1378/chest.12-1274. PMID 22910834
- [Background] Mackenzie DC, Noble VE. Assessing volume status and fluid responsiveness in the emergency department. Clin Exp Emerg Med. 2014 Dec 31;1(2):67-77. doi: 10.15441/ceem.14.040. eCollection 2014 Dec. PMID 27752556
- [Background] Levitov A, Marik PE. Echocardiographic assessment of preload responsiveness in critically ill patients. Cardiol Res Pract. 2012;2012:819696. doi: 10.1155/2012/819696. Epub 2011 Sep 12. PMID 21918726
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Blehar DJ, Glazier S, Gaspari RJ. Correlation of corrected flow time in the carotid artery with changes in intravascular volume status. J Crit Care. 2014 Aug;29(4):486-8. doi: 10.1016/j.jcrc.2014.03.025. Epub 2014 Apr 2. PMID 24930363
- [Background] Lamia B, Ochagavia A, Monnet X, Chemla D, Richard C, Teboul JL. Echocardiographic prediction of volume responsiveness in critically ill patients with spontaneously breathing activity. Intensive Care Med. 2007 Jul;33(7):1125-1132. doi: 10.1007/s00134-007-0646-7. Epub 2007 May 17. PMID 17508199
- [Background] Maizel J, Airapetian N, Lorne E, Tribouilloy C, Massy Z, Slama M. Diagnosis of central hypovolemia by using passive leg raising. Intensive Care Med. 2007 Jul;33(7):1133-1138. doi: 10.1007/s00134-007-0642-y. Epub 2007 May 17. PMID 17508202
- [Background] Stevens PM, Lamb LE. Effects of lower body negative pressure on the cardiovascular system. Am J Cardiol. 1965 Oct;16(4):506-15. doi: 10.1016/0002-9149(65)90027-5. No abstract available. PMID 5319567
- [Background] Cooke WH, Ryan KL, Convertino VA. Lower body negative pressure as a model to study progression to acute hemorrhagic shock in humans. J Appl Physiol (1985). 2004 Apr;96(4):1249-61. doi: 10.1152/japplphysiol.01155.2003. PMID 15016789
- [Background] Moore CL, Rose GA, Tayal VS, Sullivan DM, Arrowood JA, Kline JA. Determination of left ventricular function by emergency physician echocardiography of hypotensive patients. Acad Emerg Med. 2002 Mar;9(3):186-93. doi: 10.1111/j.1553-2712.2002.tb00242.x. PMID 11874773
- [Background] Moore CL, Tham ET, Samuels KJ, McNamara RL, Galante NJ, Stachenfeld N, Shelley K, Dziura J, Silverman DG. Tissue Doppler of early mitral filling correlates with simulated volume loss in healthy subjects. Acad Emerg Med. 2010 Nov;17(11):1162-8. doi: 10.1111/j.1553-2712.2010.00906.x. PMID 21175513
- [Background] Stolz LA, Mosier JM, Gross AM, Douglas MJ, Blaivas M, Adhikari S. Can emergency physicians perform common carotid Doppler flow measurements to assess volume responsiveness? West J Emerg Med. 2015 Mar;16(2):255-9. doi: 10.5811/westjem.2015.1.24301. Epub 2015 Feb 26. PMID 25834666
- [Background] Mackenzie DC, Khan NA, Blehar D, Glazier S, Chang Y, Stowell CP, Noble VE, Liteplo AS. Carotid Flow Time Changes With Volume Status in Acute Blood Loss. Ann Emerg Med. 2015 Sep;66(3):277-282.e1. doi: 10.1016/j.annemergmed.2015.04.014. Epub 2015 May 21. PMID 26003002
- [Background] Bathala L, Mehndiratta MM, Sharma VK. Transcranial doppler: Technique and common findings (Part 1). Ann Indian Acad Neurol. 2013 Apr;16(2):174-9. doi: 10.4103/0972-2327.112460. PMID 23956559
- [Background] Thomas KN, Lewis NC, Hill BG, Ainslie PN. Technical recommendations for the use of carotid duplex ultrasound for the assessment of extracranial blood flow. Am J Physiol Regul Integr Comp Physiol. 2015 Oct;309(7):R707-20. doi: 10.1152/ajpregu.00211.2015. Epub 2015 Jul 8. PMID 26157060